CLINICAL TRIAL: NCT03128827
Title: Use of Rainbow Acoustic Monitoring in Pediatric Patients - A Clinical Engineering Data Collection Protocol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Masimo Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SZMU0002
Record Dates: First submitted 2017-04-14; First posted 2017-04-25 (Actual); Last update posted 2018-10-22 (Actual); Status verified 2018-10

CONDITIONS: Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Test Subjects (Experimental): All test subjects were pediatric patients following general anesthesia who received the RAM sensor which measures respiration rate.
  Interventions: Device: RAM sensor

INTERVENTIONS:
Device: RAM sensor — Acoustic Respiration Monitor

SUMMARY:
The study will capture high resolution waveform data and numerical data from three respiratory rate methods: end tidal CO2, impedance pneumography, and bioacoustic sensing (Rainbow Acoustic Monitoring, RAM).

ELIGIBILITY:
Inclusion Criteria:

* 0 to 18 years old inclusive, male and female patients
* Only patients with written informed consent signed by parents or legal guardians will be enrolled
* In children 10 and older, patient's assent will be obtained

Exclusion Criteria:

* Patients who are unable to give their consent and/or assent
* Patients with skin abnormalities (rash, eczema, etc) at the planned application sites that would interfere with sensor, cannula or electrode applications

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 170 (Actual)
Dates: Start 2011-08-04 (Actual); Primary Completion 2015-01-20 (Actual); Study Completion 2015-07-24 (Actual)

PRIMARY OUTCOMES:
Accuracy of RAM sensor to detect respiration rate | 1-6 hours
  Accuracy will be determined by comparing the noninvasive respiratory rate measurement of the sensor to that obtained from a reference and calculating the arithmetic root mean square (Arms) error value.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Medical Center Dallas, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No